CLINICAL TRIAL: NCT05220462
Title: A Phase III Randomised, Triple-blind Controlled Superiority Trial of Remimazolam (CNS 7056), Compared to Midazolam, in Adults Having Lower Third Molar Wisdom Tooth Extraction Under Intravenous Conscious Sedation to Assess Cognitive and Motor Recovery at Normal Discharge Time
Brief Title: Remimazolam vs Midazolam Cognitive and Motor Recovery After Intravenous Conscious Sedation for Dental Extractions.
Acronym: REMIDENT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1003587
Record Dates: First submitted 2021-10-29; First posted 2022-02-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Tooth Extraction
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Experimental): White to off-white lyophilised powder, presented in a 12 mL clear glass vial with a grey bromobutyl stopper, fitted with an aluminium crimp and a blue plastic flip-off cap. Each 20 mg vial of remimazolam, will be reconstituted with sterile 0.9% NaCl solution to yield a 2.5 mg/mL solution for injection.
  An initial dose of 5mg (2mL) over 60 seconds, pausing for 90 seconds, followed by 2.5mg (1mL) over 30 seconds and waiting 30 seconds will be titrated to response end point. Subsequent doses of 2.5mg (1 mL) increments can be administered if required should the procedure take longer, or the patient recover more quickly than expected, to maintain the sedation level. Top-up doses will be administered slowly, at least 2 minutes apart. Top-up doses will be limited to a maximum of 5 doses in a 15-minute window. Additionally, a maximum dose of 40mg of remimazolam (16mL) will be set.
  Interventions: Drug: Remimazolam
- Midazolam (Active Comparator): Midazolam will be presented as a solution in a 5 mL ampoule. Each ampoule will contain 5 mg of midazolam, yielding a 1 mg/mL solution for injection.
  Dosing of midazolam was based on local formulary and standard of care / local guidance. An initial dose of 2mg (2mL) over 60 seconds, pausing for 90 seconds, followed by 1mg (1mL) over 30 seconds and waiting 30 seconds will be titrated to response end point. Subsequent doses of 1mg (1 mL) increments can be administered if required should the procedure take longer, or the patient recover more quickly than expected, to maintain the sedation level. Top-up doses will be administered slowly at least 2 minutes apart. Top-up doses will be limited to a maximum of 5 doses in a 15-minute window. Additionally, a maximum of dose of 16mg of midazolam (16mL) will be set.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam — As per Remimazolam arm
  Arms: Remimazolam
Drug: Midazolam — As per Midazolam arm
  Arms: Midazolam

SUMMARY:
The study is looking to see if a new drug (remimazolam) that is used to sedate and relax adults (aged 18-59 years) having dental treatment is better than the current drug in use (midozolam). Intravenous sedation is where a drug is injected into a patient's hand or arm. The drug stops them feeling worried, and helps them relax. After sedation, patients wait in a recovery area until they are safe to walk but the side effects of the drug can last until the next day. A new drug has been developed that has the same sedation effect and safety, but the recovery is much quicker. The investigators think that the side effects from the new drug will have worn off by the time patients are ready to leave the hospital. Patients who are coming to Guy's Hospital to have their wisdom tooth extracted under sedation will be asked if they want to be included in the research. Patients will be randomised to receive either remimazolam of standard of care midazolam. The sedation and dental treatment will be carried out in the normal way.

The patients will be asked to do will be some questionnaires and some tests which are as follows:

1. Patients are asked to listen to some words and repeat them back. This tests how well they can remember new information
2. Reaction test - Patients are asked to rest their fingers on a keypad and move their fingers when lights come on above them. This tests how quick their reactions are.
3. Symbol test- Patients are asked to draw small shapes that are linked to numbers. This tests how well they can process information.
4. Standing test- Patients are asked to stand on a platform that measures how much they are swaying back and forth. This tests how stable they are to walk.

By testing people before and after the sedation the investigators can see how they recovered and compare the two drugs. The research will take place during the day case visit and involve 2 x 30 mins research assessments (before sedation and post sedation). After the post-sedation tests, participants will be discharged, followed by a telephone review 3-10 days post procedure.

DETAILED DESCRIPTION:
This study will be performed as a prospective, randomised, triple blind, active controlled, parallel group, single centre study design assessing enhanced cognitive recovery in patients having third molar wisdom tooth extraction under intravenous conscious sedation with remimazolam. An active control group has been chosen using intravenous midazolam which is the current standard of care in Dentistry. 128 patients will be randomised, of which n=64 will receive remimazolam, and n=64 in the midazolam group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to have mandibular third molar removal with intravenous conscious sedation.
* Male and female patients, aged ≥18 to ≤59 years old.
* American Society of Anesthesiologists (ASA-PS) grade I or II.
* English as their first or main language for 5+ years. The primary outcome measure (HVLT) is a cognitive test to remember English words and validated on this basis.
* A patient who has given informed written consent for inclusion to the study.
* Patients who are willing and able to comply with study requirements.

Exclusion Criteria:

* Any surgical risk factor which, in the opinion of the study surgeon, can lead to increased procedure complexity (for example high risk of inferior alveolar nerve damage)
* A known sensitivity to benzodiazepines or a medical condition such that these agents are contraindicated as per the SmPC, for example unstable myasthenia gravis, hepatic impairment, acute respiratory depression, and severe respiratory failure.
* Any neurological deficit where cognitive tests will be impaired (for example dementia).
* A patient with known difficult airway/ mask ventilation or who has increased risk factors recorded by the clinical team at assessment.
* A patient who reports hypersensitive gag reflex.
* Body mass index >34.9 kg/m or weight <50kg or >130kg.
* Dental or needle phobia identified by a modified dental anxiety score ≥19 (MDAS questionnaire).
* High Hospital Anxiety and Depression Score (HADS) >12.
* Chronic use of benzodiazepines or opioids for any indication.
* Use of medications known to interact with IMP or comparator as listed in the SmPC.
* All female patients with a positive urine pregnancy test within 8 hours before IMP administration. Female patients who are permanently sterile are not required to have a urine test. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
* Lactating female patients currently breastfeeding.
* Patients who self-report illicit drug use in the last 4 weeks. Patients who self-report alcohol abuse (AUDIT-C Scores > 7) or history of abuse within the past 5 years.
* Patients who self-report a history of illicit drug abuse within the past 5 years or any history of benzodiazepine dependence.
* Inclusion in a study of an IMP in the previous 4 weeks or less than seven half-lives (whichever is the longer).
* Hypersensitivity to the IMP or to any of the excipients.
* Patients who are unable to stand unassisted.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test Revised (HVLT-R) | On day 1. At time T60 (60 minutes after last dose of IMP)
  The sum of the correct responses in the three learning trials (total recall) following last dose administration of remimazolam or midazolam.

SECONDARY OUTCOMES:
Cognitive and Motor Testing | Baseline and 60 minutes (T60)
  Proportion of patients returning to within 1 standard error (SE) of pre-dose cognitive and motor testing.
Digit Symbol Substitution Test (DSST) | Baseline and 60 minutes (T60)
  Number of items completed on the digit symbol substitution test (DSST) at baseline and 60 minutes following last dose administration of remimazolam or midazolam
Balance Board | Baseline and 60 minutes (T60)
  Scores on the scales for assessment and rating of ataxia (balance board) at baseline and 60 minutes following last dose administration of remimazolam or midazolam
MOART Device | Baseline and 60 minutes (T60)
  Scores on the reaction time measured on a MOART device by choice reaction time (with Go/No Go) at baseline and 60 minutes following last dose administration of remimazolam or midazolam
Start of Procedure | Time-to-event from IMP administration to start of procedure recorded in minutes between 0 minutes and 20 minutes
  The time to start of procedure (local anaesthetic injection) after administration of the first dose of study medication.
Fully Alert After End of Procedure - Modified Observer's Assessment of Alertness/Sedation (MOAA/S) | On day 1. Time in minutes between 0 and 90 minutes after defined procedure end.
  The times to fully alert (first of three Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores of 5 after the end of the procedure (surgical "time out").
Fully Alert After Last Injection of Study Drug - Modified Observer's Assessment of Alertness/Sedation (MOAA/S) | On day 1. Time in minutes between 0 and 90 minutes after last dose of IMP.
  The times to fully alert (first of three Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores of 5 after the last injection of study drug.
Ready for Discharge After End of Procedure | On day 1. Time in minutes between 0 and 90 minutes after defined procedure end.
  The times to initial recovery and ready for discharge (passed walk test) after the end of the procedure (surgical "time out").
Ready for Discharge After Last Injection of Study Drug | On day 1. Time in minutes between 0 and 90 minutes after last dose of IMP
  The times to initial recovery and ready for discharge (passed walk test) after the last injection of study drug .
Dental Sedation Teachers Group (DSTG) Score | On day 1. Assessed up to 60 minutes after end of procedure (surgical "time out")
  The overall co-operation score given by the surgical team (DSTG score).
  The scale is 1 (good) to 4 (impossible), with 1 being the better outcome.
Visual Analogue Score (VAS) | On day 1. Assessed up to 5 minutes after dosing IMP
  Occurrence of pain on injection at application of study medication (VAS).
  The scale is 1-10, with 1 being the better outcome.
The Patient Satisfaction Score | On day 1 at discharge and repeated on review phone call (minimum on day 3, up to day 10 after procedure)
  The patient satisfaction score
  The questionnaire has multiple questions, which the patient will score from 0-10. 10 is the better outcome.
Requirement for Flumazenil during the Procedure or to Aid Recovery. | During procedure
  The requirement for flumazenil during the procedure or to aid recovery.
Inadequate Sedation | During procedure
  The procedure failure rate due to inadequate sedation at the maximum dose / top-up rate
Comparison of Safety Measures - Hypoxia | During Procedure
  Comparison of safety measures - hypoxia (SpO2).
Comparison of Safety Measures - Airway Manoeuvres | During Procedure
  Comparison of safety measures - use of airway manoeuvres.
Comparison of Safety Measures - Heart Rate | During Procedure
  Comparison safety measures - bradycardia & tachycardia (pulse).
Comparison of Safety Measures - Blood Pressure | During Procedure
  Comparison of safety measures - hypotension and hypertension (NIBP).

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Kerr, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD